CLINICAL TRIAL: NCT02336737
Title: A Pivotal, Prospective, Open-Label, Multicenter Paired Comparison Study Of SentiMag/SiennaXP And The Standard Of Care In Patients With Breast Cancer Who Are Undergoing Lymph Node Mapping As Part Of A Sentinel Node Biopsy Procedure
Brief Title: SentiMag® Intraoperative Comparison in Breast Cancer
Acronym: SentiMagIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endomagnetics Inc (Industry)
Collaborators: Regulatory and Clinical Research Institute Inc (Other)
Responsible Party: Sponsor
Organization: Endomagnetics Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: US-001
Record Dates: First submitted 2015-01-07; First posted 2015-01-13 (Estimated); Results first posted 2020-11-03 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Breast Cancer
Keywords: breast cancer; sentinel lymph node biopsy
MeSH Terms: conditions — Breast Neoplasms | interventions — Technetium Tc 99m Sulfur Colloid; Radioisotopes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SiennaXP injection (Experimental): Single injection of SiennaXP in addition to comparator single dose of radioisotope (Technetium Tc99m Sulfur Colloid) and single dose of isosulfan blue dye.
  Lymph node localization using the SentiMag handheld intraoperative localization system in addition to localization with standard of care handheld gamma probe.
  Interventions: Device: SiennaXP; Drug: Technetium Tc99m Sulfur Colloid; Drug: Isosulfan blue dye

INTERVENTIONS:
Device: SiennaXP — Sub-cutaneous injection of SiennaXP magnetic marker, followed by lymph node localization using the SentiMag handheld magnetic probe
Drug: Technetium Tc99m Sulfur Colloid — Injection of a single dose of radioisotope (Technetium Tc99m Sulfur Colloid)
  Other Names: Radioisotope
Drug: Isosulfan blue dye — Injection of a single dose of isosulfan blue dye
  Other Names: Blue dye

SUMMARY:
The purpose of this pivotal study is to provide prospective evidence that the SentiMag®/SiennaXP® is safe and non-inferior to the current standard of care for lymph node localization in patients with breast cancer as part of a sentinel lymph node biopsy (SLNB) procedure and to summarize measures of product safety and performance.

DETAILED DESCRIPTION:
This is a pivotal, prospective, open label, multicenter, paired comparison of the SentiMag® and SiennaXP® magnetic sentinel node localization system with the standard of care (radioisotope with blue dye) for lymph node localization in the detection of lymph nodes in patients with breast cancer undergoing a sentinel lymph node biopsy. The trial is designed to provide powered evidence that the lymph node detection rate of the SentiMag® and SiennaXP® system is non-inferior to the standard of care in patients with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of primary breast cancer or subjects with pure ductal carcinoma in situ (DCIS).
* Subjects scheduled for surgical intervention, with a sentinel lymph node biopsy procedure being a part of the surgical plan.
* Subjects aged 18 years or more at the time of consent.
* Subjects with an ECOG (Eastern Cooperative Oncology Group) performance status of Grade 0 - 2.
* Subject has a clinical negative node status (i.e. T0-3, N0, M0).

Exclusion Criteria:

* The subject is pregnant or lactating.
* The subject has clinical or radiological evidence of metastatic cancer including palpably abnormal or enlarged lymph nodes.
* The subject has a known hypersensitivity to Isosulfan Blue Dye.
* The subject has participated in another investigational drug study within 30 days of scheduled surgery.
* Subject has had either a) previous axilla surgery, b) reduction mammoplasty, or c) lymphatic function that is impaired in the surgeon's judgment.
* Subject has had preoperative radiation therapy to the affected breast or axilla.
* Subject has received a Feraheme® (ferumoxytol) Injection within the past 6 months.
* Subject has intolerance or hypersensitivity to iron or dextran compounds or to SiennaXP.
* Subject has an iron overload disease.
* Subject has pacemaker or other implantable device in the chest wall.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Alvarado, MD, Principal Investigator — University of CA, San Francisco Carol Franc Buck Breast Care, Dept of Surgery
Locations (6):
- United States (6):
  - University of California San Diego Moores Cancer Center, La Jolla, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCSF Carol Franc Buck Breast Care Center, San Francisco, California
  - Coordinated Health Breast Care Specialists, Allentown, Pennsylvania
  - Dallas Surgical Group, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Background] Douek M, Klaase J, Monypenny I, Kothari A, Zechmeister K, Brown D, Wyld L, Drew P, Garmo H, Agbaje O, Pankhurst Q, Anninga B, Grootendorst M, Ten Haken B, Hall-Craggs MA, Purushotham A, Pinder S; SentiMAG Trialists Group. Sentinel node biopsy using a magnetic tracer versus standard technique: the SentiMAG Multicentre Trial. Ann Surg Oncol. 2014 Apr;21(4):1237-45. doi: 10.1245/s10434-013-3379-6. Epub 2013 Dec 10. PMID 24322530
- [Background] Thill M, Kurylcio A, Welter R, van Haasteren V, Grosse B, Berclaz G, Polkowski W, Hauser N. The Central-European SentiMag study: sentinel lymph node biopsy with superparamagnetic iron oxide (SPIO) vs. radioisotope. Breast. 2014 Apr;23(2):175-9. doi: 10.1016/j.breast.2014.01.004. Epub 2014 Jan 29. PMID 24484967

RESULTS

PARTICIPANT FLOW:
Groups:
- SiennaXP Injection: Single injection of SiennaXP in addition to comparator single dose of radioisotope (Technetium Tc99m Sulfur Colloid) and single dose of isosulfan blue dye.
  Lymph node localization using the SentiMag handheld intraoperative localization system in addition to localization with standard of care handheld gamma probe.
  SiennaXP: Sub-cutaneous injection of SiennaXP magnetic marker, followed by lymph node localization using the SentiMag handheld magnetic probe
  Technetium Tc99m Sulfur Colloid: Injection of a single dose of radioisotope (Technetium Tc99m Sulfur Colloid)
  Isosulfan blue dye: Injection of a single dose of isosulfan blue dye
Period: Overall Study
Arm/Group | SiennaXP Injection
Started | 160
Completed | 147
Not Completed | 13
Not completed — Withdrawal by Subject | 5
Not completed — Physician Decision | 8

BASELINE CHARACTERISTICS:
Units Other Than Participants: Sentinel Lymph Nodes (SLN)
Groups:
- SiennaXP Injection: Single injection of SiennaXP in addition to comparator single dose of radioisotope (Technetium Tc99m Sulfur Colloid) and single dose of isosulfan blue dye.
  Lymph node localization using the SentiMag handheld intraoperative localization system in addition to localization with standard of care handheld gamma probe.
  SiennaXP: Sub-cutaneous injection of SiennaXP magnetic marker, followed by lymph node localization using the SentiMag handheld magnetic probe
  Technetium Tc99m Sulfur Colloid: Injection of a single dose of radioisotope (Technetium Tc99m Sulfur Colloid)
Arm/Group | SiennaXP Injection
Number analyzed (Participants) | 147
Number analyzed (Sentinel Lymph Nodes (SLN)) | 369
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 90
  >=65 years | 57
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.1 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex of study subject was recorded
  Participants
    Female | 147
    Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Study subjects self-reported their ethnicity
  Participants
    Hispanic or Latino | 17
    Not Hispanic or Latino | 130
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Study subjects self reported their race
  Participants
    American Indian or Alaska Native | 0
    Asian | 7
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 11
    White | 121
    More than one race | 0
    Unknown or Not Reported | 8
Region of Enrollment [Number; unit: subjects] — Country where study was being conducted
  subjects
    United States | 147

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Detected Lymph Nodes
Description: The proportion of lymph nodes detected intraoperatively by SentiMag and SiennaXP in relation the proportion of lymph nodes detected by the combination of Technetium Sulfur Colloid and Isosulfan blue dye
Time Frame: During surgical procedure <1 hour
Population: 146/147 were evaluated for the primary objective. One (1) subject had missing data and therefore was not included in the primary endpoint analysis
Measure: Count of Participants; unit: Participants
Arm/Group | SiennaXP Injection
Number analyzed (Participants) | 146
Participants | 145

2. Primary Outcome: Safety of SiennaXP and SentiMag® as Indicated by Adverse Events and Serious Adverse Events and Their Relatedness to the Detection Method or Procedure.
Description: Number of Participants with Adverse Events relating to Sienna XP Injection
Time Frame: 3-6 weeks
Population: Number of subjects experiencing Sienna XP injection-related adverse events from enrollment through subject exit or completion
Measure: Count of Participants; unit: Participants
Arm/Group | SiennaXP Injection
Number analyzed (Participants) | 160
Participants | 20

3. Secondary Outcome: Nodal Concordance: Number of Nodes Identified by Both Test and Control Out of Nodes Identified by Control
Description: The number of nodes identified by both SiennaXP and Control out of nodes identified by Control
Time Frame: Intraoperative <1 hour
Measure: Number (95% Confidence Interval); unit: percentage of concordance
Arm/Group | SiennaXP Injection
Number analyzed (Participants) | 147
percentage of concordance | 94.5 [92.1 to 96.9]

4. Secondary Outcome: Number of Participants With Lymph Nodes Detected by Combined Radioisotope,Blue Dye and Magnetic Technique
Description: The per patient detection rate for a combination of all methods (magnetic, combined radioisotope and blue dye; radioisotope alone; blue dye alone)
Time Frame: Intraoperative <1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | SiennaXP Injection
Number analyzed (Participants) | 146
Participants | 145

ADVERSE EVENTS:
Arm/Group | SiennaXP Injection
All-Cause Mortality (participants affected / at risk) | 0/147
Serious Adverse Events (participants affected / at risk) | 0/147
Other Adverse Events (participants affected / at risk) | 23/147
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SiennaXP Injection (N=147)
Breast discolouration/hyperpigmentation (Skin and subcutaneous tissue disorders) | 23 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No